CLINICAL TRIAL: NCT03538834
Title: The Effects of a Daily Intake of Cod Residual Material Meal for 8 Weeks on Serum Lipids and Fatty Acids, Glucose Regulation and Body Composition in Lean, Active Adults: A Randomized Controlled Trial.
Brief Title: The Effects of Dietary Intake of Cod Residual Material Meal on Lipid Regulation, Glucose Regulation and Body Composition in Physically Active Adults
Acronym: COD2016
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other); K. Halstensen AS (Unknown); Regional Research Fund Western Norway (Unknown); Nofima (Other)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, Researcher, PhD, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2015/75 part 2
Record Dates: First submitted 2018-05-14; First posted 2018-05-29 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Physical Activity; Healthy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cod meal from residual material (Experimental): Dietary supplement: cod meal from residual material, 8 g protein daily for 8 weeks
  Interventions: Dietary Supplement: Cod meal from residual material
- Control (Placebo Comparator): Control group receive tablet containing fillers and no protein
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Cod meal from residual material — Cod meal from residual material, 8 g protein daily for 8 weeks
  Arms: Cod meal from residual material
Dietary Supplement: Control — Placebo
  Arms: Control

SUMMARY:
A high intake of fish is associated with positive health effects, including prevention and treatment of chronic non-communicable diseases, such as cardiovascular diseases (CVDs) and type 2 diabetes. These health effects have traditionally been attributed to the omega-3 fatty acids in fatty fish, but recent studies have suggested that also fish proteins may improve biomarkers of metabolic disease. Intake of cod fillet have previously shown beneficial effects on blood lipids, glucose regulation and body composition in adults with overweight or obesity. Health effect of cod residual material from fillet production (i.e., head, backbone, skin, cutoffs and entrails) have so far not been investigated, but residuals from other fish species have shown promising effects on glucose regulation in rats. The main aim of the current study is to investigate the effects of cod residual meal on serum lipids and glucose regulation in healthy, physically active adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 18.5 kg/m2
* Fasting blood glucose ≤7 mmol/L
* Physically active
* Percent body fat, 5-25 % for men and 12-35 % for women

Exclusion Criteria:

* Allergies towards fish, milk, egg, gluten
* Tobacco use > 10 cigarettes (or snus) per day
* Diseases affecting the heart, intestinal function, kidney function or insulin secretion
* Medications targeting cholesterol -or glucose metabolism, hypertension
* Use of dietary supplements
* Pregnancy or lactation

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Lipid metabolism | 8 weeks
  Lipids will be measured in fasting serum samples

SECONDARY OUTCOMES:
Biomarkers related to glucose regulation | 8 weeks
  Glucose, insulin and GLP-1 and will be measured in serum/plasma sampled in fasting and postprandial conditions
Body composition | 8 weeks
  Percent body fat will be measured using bioimpedance

CONTACTS AND LOCATIONS:
Locations (1):
- Oddrun Anita Gudbrandsen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vikoren LA, Nygard OK, Lied E, Rostrup E, Gudbrandsen OA. A randomised study on the effects of fish protein supplement on glucose tolerance, lipids and body composition in overweight adults. Br J Nutr. 2013 Feb 28;109(4):648-57. doi: 10.1017/S0007114512001717. Epub 2012 May 31. PMID 22647247
- [Background] Drotningsvik A, Mjos SA, Pampanin DM, Slizyte R, Carvajal A, Remman T, Hogoy I, Gudbrandsen OA. Dietary fish protein hydrolysates containing bioactive motifs affect serum and adipose tissue fatty acid compositions, serum lipids, postprandial glucose regulation and growth in obese Zucker fa/fa rats. Br J Nutr. 2016 Oct;116(8):1336-1345. doi: 10.1017/S0007114516003548. Epub 2016 Oct 18. PMID 27751188
- [Background] Vildmyren I, Cao HJV, Haug LB, Valand IU, Eng O, Oterhals A, Austgulen MH, Halstensen A, Mellgren G, Gudbrandsen OA. Daily Intake of Protein from Cod Residual Material Lowers Serum Concentrations of Nonesterified Fatty Acids in Overweight Healthy Adults: A Randomized Double-Blind Pilot Study. Mar Drugs. 2018 Jun 5;16(6):197. doi: 10.3390/md16060197. PMID 29874805